CLINICAL TRIAL: NCT00487942
Title: A 4-Week, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dosage Study to Evaluate the Efficacy and Safety of Armodafinil as Adjunctive Therapy in Adults With Cognitive Deficits Associated With Schizophrenia
Brief Title: Efficacy and Safety of Armodafinil as Adjunctive Therapy in Schizophrenic Adults With Cognitive Deficits
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor's Medical Expert, Cephalon
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/2033/SZ/US
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 50 mg/day armodafinil (Active Comparator): Armodafinil or placebo was provided in 50 mg tablet form and subjects were instructed to take 4 tablets orally once daily in the morning. Subjects randomized to the 50 mg/day armodafinil treatment arm for the double-blind treatment period of the study took one 50 mg armodafinil tablet plus three placebo tablets each morning.
  Interventions: Drug: armodafinil
- 100 mg/day armodafinil (Active Comparator): Armodafinil or placebo was provided in 50 mg tablet form and subjects were instructed to take 4 tablets orally once daily in the morning. Subjects randomized to the 100 mg/day armodafinil treatment arm for the double-blind treatment period of the study took two 50 mg armodafinil tablets plus two placebo tablets each morning. Subjects began taking 50 mg/day and then titrated to 100 mg/day on Day 2 of the first week of the double-blind treatment period.
  Interventions: Drug: armodafinil
- 200 mg/day armodafinil (Active Comparator): Armodafinil or placebo was provided in 50 mg tablet form and subjects were instructed to take 4 tablets orally once daily in the morning. Subjects randomized to the 200 mg/day armodafinil treatment arm for the double-blind treatment period of the study took four 50 mg armodafinil tablet and no placebo tablets each morning. Subjects were titrated to this dose by starting treatment at 50 mg/day (1 tablet) and increasing by 50 mg increments on days 2, 4, and 6 until they were taking 200 mg/day.
  Interventions: Drug: armodafinil
- Placebo (Placebo Comparator): Armodafinil or placebo was provided in 50 mg tablet form and subjects were instructed to take 4 tablets orally once daily in the morning. Subjects randomized to the placebo treatment arm for the double-blind treatment period of the study took four placebo tablets and no armodafinil tablets each morning.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil — 50 mg/day armodafinil
  Arms: 50 mg/day armodafinil
Drug: armodafinil — 100 mg/day armodafinil
  Arms: 100 mg/day armodafinil
Drug: armodafinil — 200 mg/day armodafinil
  Arms: 200 mg/day armodafinil
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate if adjunctive armodafinil treatment can improve the cognitive deficits in patients with schizophrenia

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has a diagnosis of schizophrenia according to the DSM-IV-TR criteria as determined by the SCID and has been clinically stable in a nonacute phase of their illness for at least 8 weeks prior to the baseline visit.
* The patient has received treatment with olanzapine, oral risperidone, or paliperidone for schizophrenia for at least 6 weeks prior to the screening visit and has been on a stable dose of olanzapine, oral risperidone, or paliperidone for at least 4 weeks prior to the screening visit. The patient is prepared to remain at these stable dosages for the duration of the study.
* The patient is a man or woman 18 through 60 years of age.
* The patient is in good health (except for the diagnosis of schizophrenia) as judged by the investigator on the basis of medical and psychiatric history, medical examination, ECG, serum chemistry, hematology, and urinalysis.
* Women of childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* The patient must be willing and able to comply with study restrictions, to remain at the clinic for the required duration during the study period, and to return to the clinic for the follow-up evaluation as specified in this protocol.

Key Exclusion Criteria:

* The patient has any Axis I disorder, including schizoaffective disorder and sleep disorders, apart from schizophrenia, and nicotine dependence.
* The patient has tardive dyskinesia or any other clinically significant movement disorder.
* The patient has any clinically significant uncontrolled medical (including illnesses related to the cardiovascular, renal, or hepatic systems) or surgical condition.
* The patient has previously received modafinil or armodafinil, or the patient has a known sensitivity to any ingredients in the study drug tablets.
* The patient is a pregnant or lactating woman. (Any woman becoming pregnant during the study will be withdrawn from the study.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Collaborative NeuroScience Network, Garden Grove, California
  - Synergy Clinical Research, National City, California
  - California Clinical Trials, Paramount, California
  - CNRI-Los Angeles, LLC, Pico Rivera, California
  - CNRI-San Diego, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Atlanta Center for Clinical Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Department of Psychiatry - DUMC, Durham, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - University Hills Clinical Research, Irving, Texas

REFERENCES:
- [Derived] Kane JM, D'Souza DC, Patkar AA, Youakim JM, Tiller JM, Yang R, Keefe RS. Armodafinil as adjunctive therapy in adults with cognitive deficits associated with schizophrenia: a 4-week, double-blind, placebo-controlled study. J Clin Psychiatry. 2010 Nov;71(11):1475-81. doi: 10.4088/JCP.09m05950gry. Epub 2010 Aug 24. PMID 20816042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven centers in the United States (US). First participant enrolled: July 2007 / Last participant last visit: December 2007
Pre-assignment Details: The study consisted of a screening period of at least 1 week, a 4 week double blind treatment period, and a 1 week follow up period. Of the 60 patients enrolled, 59 patients received at least 1 dose of study drug and were evaluated for safety; 1 patient who was assigned to receive placebo withdrew before taking any study drug.
Groups:
- Armodafinil 50 mg/Day: Patients took 4 tablets orally, once daily in the morning. The 4 tablets consumed consisted of one 50 mg active tablet of armodafinil and three placebo tablets. Patients remained at their randomized dosage for the duration of the study.
- Armodafinil 100 mg/Day: Patients took 4 tablets orally, once daily in the morning. Treatment with study drug began at 50 mg/day (one 50 mg armodafinil tablet and three placebo tablets) and was titrated in a 50 mg increment to the randomized dosage of 100 mg/day (two 50 mg armodafinil tablets and two placebo tablets) on day 2. Patients remained at their randomized dosage for the duration of the study.
- Armodafinil 200 mg/Day: Patients took 4 tablets orally, once daily in the morning. Treatment with study drug began at 50 mg/day (one 50 mg armodafinil tablet and three placebo tablets) and was titrated in 50 mg increments (an additional 50 mg armodafinil tablet and one less placebo tablet), as appropriate, on days 2, 4, and 6 to the randomized dosage of 200 mg/day (four 50 mg armodafinil tablets and no placebo tablets). Patients remained at their randomized dosage for the duration of the study.
- Placebo: Placebo tablets matching the 50 mg armodafinil tablet were used in a manner identical to that of the armodafinil tablets for those patients administered placebo during the double blind treatment period.
Period: Overall Study
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Started | 15 | 15 | 15 | 15 (One subject randomized to placebo discontinued prior to receiving any study drug, leaving 14.)
Completed | 12 | 12 | 12 | 13
Not Completed | 3 | 3 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.9 (10.88) | 40.4 (9.58) | 41.4 (9.78) | 46.0 (7.80) | 43.2 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 3 | 16
  Male | 11 | 10 | 11 | 12 | 44
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Last Observation After Baseline in Composite Score on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The composite score combines the individual scores of the 10 tests and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represents the change from baseline to last observation after baseline in Composite T-Score.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had at least 1 MATRICS efficacy assessment after baseline. If any part of the composite score was missing then the composite score was set to missing. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 13 | 11 | 13
Units on a scale | 1.9 (6.22) | 2.8 (7.98) | 2.9 (4.72) | 2.2 (5.06)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil treatment in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the composite score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; ANCOVA — Inferential statistics were not performed; Effect size = -0.04, 95% CI 2-sided [-0.81 to 0.73]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA — Inferential statistics were not performed; Effect size = 0.09, 95% CI 2-sided [-0.68 to 0.86]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA — Inferential statistics were not performed; Effect size = 0.15, 95% CI 2-sided [-0.66 to 0.95]

2. Secondary Outcome: Change From Baseline to Week 4 in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery Composite Score
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The composite score combines the individual scores of the 10 tests and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in composite T-score from baseline to 4 weeks.
Time Frame: Baseline and 4 weeks
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had a MATRICS efficacy assessment at baseline and at Week 4. If any part of the composite score was missing then the composite score was set to missing. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12
Units on a scale | 2.2 (6.13) | 3.9 (5.99) | 2.9 (4.72) | 2.1 (5.28)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.02, 95% CI 2-sided [-0.80 to 0.83]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.31, 95% CI 2-sided [-0.51 to 1.14]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.16, 95% CI 2-sided [-0.66 to 0.98]

3. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Speed of Processing Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in Processing Speed Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline 4 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had at least 1 MATRICS efficacy assessment after baseline. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 3.0 (8.81) | 0.0 (10.42) | 5.0 (9.14) | 0.9 (6.95)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.25, 95% CI 2-sided [-0.51 to 1.01]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.10, 95% CI 2-sided [-0.86 to 0.66]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.49, 95% CI 2-sided [-0.31 to 1.28]

4. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Attention/Vigilance Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument containing 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in Attention/Vigilance Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 12 | 13
Units on a scale | 0.4 (10.89) | 3.7 (5.02) | 1.8 (6.51) | 3.0 (6.56)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.27, 95% CI 2-sided [-1.03 to 0.48]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential Statistics were not performed; Effect Size = 0.11, 95% CI 2-sided [-0.65 to 0.88]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.18, 95% CI 2-sided [-0.97 to 0.60]

5. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Working Memory Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in Working Memory Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 2.3 (6.51) | 4.3 (6.02) | 3.5 (10.41) | 4.4 (6.33)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.32, 95% CI 2-sided [-1.08 to 0.44]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential Statistics were not performed; Effect Size = -0.02, 95% CI 2-sided [-0.77 to 0.74]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.10, 95% CI 2-sided [-0.89 to 0.68]

6. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Verbal Learning Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in Verbal Learning Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -1.2 (6.31) | -0.8 (4.49) | 0.8 (6.31) | -2.2 (5.93)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.15, 95% CI 2-sided [-0.61 to 0.90]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.25, 95% CI 2-sided [-0.50 to 1.01]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.46, 95% CI 2-sided [-0.34 to 1.25]

7. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Visual Learning Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, where the mean is 50 and a standard deviation is 10 for the composite. The data here represent the mean change in Visual Learning Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 14 | 11 | 13
Units on a scale | 4.3 (9.55) | 3.9 (12.84) | 1.3 (8.76) | 0.2 (8.15)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.45, 95% CI 2-sided [-0.33 to 1.23]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.34, 95% CI 2-sided [-0.42 to 1.10]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.13, 95% CI 2-sided [-0.68 to 0.93]

8. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Reasoning and Problem Solving Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument containing 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10) for the composite. The data here represent the mean change in Reasoning and Problem Solving Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 1.6 (4.31) | -0.4 (5.60) | -0.3 (8.36) | -0.2 (4.63)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.39, 95% CI 2-sided [-0.37 to 1.15]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.05, 95% CI 2-sided [-0.81 to 0.70]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.01, 95% CI 2-sided [-0.80 to 0.77]

9. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Social Cognition Domain of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Domain score combines the individual test scores of the Domain and scores them on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10) for the composite. The data here represent the mean change in Social Cognition Domain T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -3.1 (6.93) | -1.3 (8.20) | 3.6 (8.26) | 3.8 (6.62)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.99, 95% CI 2-sided [-1.79 to -0.19]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.66, 95% CI 2-sided [-1.44 to 0.11]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.03, 95% CI 2-sided [-0.82 to 0.75]

10. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Trail Making Test of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Trail Making Test is a component of the Speed of Processing Domain scored on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10). The data here represent the mean change in Trail Making Test T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 4.2 (13.15) | -0.2 (11.76) | 9.2 (15.43) | -1.0 (7.80)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.46, 95% CI 2-sided [-0.30 to 1.23]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.08, 95% CI 2-sided [-0.68 to 0.83]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.81, 95% CI 2-sided [-0.00 to 1.63]

11. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Brief Assessment of Cognition in Schizophrenia: Symbol Coding (BASC SC) Test of the MATRICS Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The BASC SC Test is a component of the Speed of Processing Domain scored on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10). The data here represent the mean change in BASC SC Test T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 0.6 (9.14) | -0.4 (11.26) | 2.4 (7.93) | 4.0 (7.25)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.39, 95% CI 2-sided [-1.16 to 0.37]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.45, 95% CI 2-sided [-1.21 to 0.31]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.20, 95% CI 2-sided [-0.99 to 0.58]

12. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Fluency Test of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The Fluency Test is a component of the Speed of Processing Domain scored on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10). The data here represent the mean change in Fluency Test T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 2.2 (7.81) | 0.8 (7.83) | -0.5 (4.68) | -1.4 (7.12)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.47, 95% CI 2-sided [-0.30 to 1.23]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = 0.28, 95% CI 2-sided [-0.48 to 1.04]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.14, 95% CI 2-sided [-0.64 to 0.93]

13. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Wechsler Memory Scale: Spatial Span (WMS-III SS) Test of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The WMS-III SS is a component of the Working Memory Domain scored on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10). The data here represent the mean change in WMS-III SS T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 0.7 (8.47) | 4.7 (7.21) | 2.9 (8.08) | 2.5 (5.67)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.23, 95% CI 2-sided [-0.99 to 0.52]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.34, 95% CI 2-sided [-0.42 to 1.10]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.06, 95% CI 2-sided [-0.72 to 0.85]

14. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Letter-Number Span (LNS) Test of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
Description: The MATRICS Consensus Cognitive Battery is an instrument that contains 10 tests to measure cognitive performance in 7 cognitive domains: speed processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The LNS is a component of the Working Memory Domain scored on a normative scale to derive a T-score, (mean is 50 and standard deviation is 10). The data here represent the mean change in LNS T-score from baseline to last observation after baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 3.1 (6.32) | 2.1 (6.16) | 3.1 (9.63) | 4.5 (6.79)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.20, 95% CI 2-sided [-0.95 to 0.56]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.35, 95% CI 2-sided [-1.11 to 0.41]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.16, 95% CI 2-sided [-0.95 to 0.62]

15. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Wisconsin Card Sort Test (WCST) - Number of Perseverative Errors
Description: WCST is an instrument administered electronically to assess abstract reasoning and ability to alter problem solving strategies. Patients are given 64 response cards and 4 stimulus cards and asked to match each stimulus card to 1 pile of response cards. The patient is not told how to match the cards, only "right" or "wrong" to each placement. Examiner may change matching rules during the test. Perseveration errors occur when subject repeats the same error no matter how many times they are told the placement is wrong. The change from baseline in number of perseveration errors was assessed.
Time Frame: 4 weeks (or last observation after baseline)
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had at least 1 efficacy assessment after baseline. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 12 | 12
Errors | 1.6 (5.35) | -8.0 (12.79) | -2.2 (11.75) | -1.9 (7.77)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.51, 95% CI 2-sided [-1.30 to 0.27]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.55, 95% CI 2-sided [-0.25 to 1.35]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.02, 95% CI 2-sided [-0.78 to 0.82]

16. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Wisconsin Card Sort Test (WCST) - Consecutive Responses on the Final Category
Description: WCST is an instrument administered electronically to assess abstract reasoning and ability to alter problem solving strategies. Patients are given 64 response cards and 4 stimulus cards and asked to match each stimulus card to 1 pile of response cards. The patient is not told how to match the cards, only "right" or "wrong" to each placement. Examiner may change matching rules (sorting categories) during the test at which time the subject must alter their sorting category. The change from baseline in number of consecutive responses on the final category was assessed.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Responses
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 12 | 12
Responses | -1.6 (2.98) | -0.5 (4.46) | 0.3 (2.64) | 0.7 (3.80)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.64, 95% CI 2-sided [-1.43 to 0.15]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect Size = -0.26, 95% CI 2-sided [-1.05 to 0.53]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.10, 95% CI 2-sided [-0.90 to 0.70]

17. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Wisconsin Card Sort Test (WCST) - Categories Completed
Description: WCST is an instrument administered electronically to assess abstract reasoning and ability to alter problem solving strategies. Patients are given 64 response cards and 4 stimulus cards and asked to match each stimulus card to 1 pile of response cards. The patient is not told how to match the cards, only "right" or "wrong" to each placement. Examiner may change matching rules (sorting categories) during the test at which time the subject must alter their sorting category. The change from baseline in number of sorting categories achieved was assessed.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Categories Completed
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 12 | 12
Categories Completed | 0.0 (1.36) | 0.5 (1.85) | -0.3 (1.66) | 0.2 (0.72)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.15, 95% CI 2-sided [-0.92 to 0.63]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.25, 95% CI 2-sided [-0.54 to 1.04]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.31, 95% CI 2-sided [-1.12 to 0.49]

18. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Trails B Test
Description: Trail B is an instrument designed to assess set shifting. The patient was given a paper with numbers and letters on it and asked to connect them in an alternating manner (eg. 1-A-2-B-3C). The time required for the patient to complete the test was recorded. The change from Baseline to last observation following Baseline in the time necessary to complete the test is presented here.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 13 | 10 | 13
Minutes | -8.7 (41.45) | 17.5 (56.31) | -20.8 (61.93) | -27.6 (40.92)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil treatment in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the Trails B Test score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics not performed; Effect size = -0.44, 95% CI 2-sided [-1.22 to 0.33]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Inferential statistics not performed; Effect size = -0.89, 95% CI 2-sided [-1.69 to -0.08]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Inferential statistics not performed; Effect size = -0.13, 95% CI 2-sided [-0.95 to 0.70]

19. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Median Value for Actigraphy Data of Average Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in average activity per epoch (counts/epoch).
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had a baseline and at least one post-baseline assessment by actigraphy
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -17.6 (25.81) | -0.7 (27.33) | 4.2 (27.77) | 0.8 (32.98)

20. Secondary Outcome: Change From Baseline to Week 1 in the Median Value for Actigraphy Data of Average Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in average activity per epoch (counts/epoch)to Week 1.
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -2.3 (43.02) | 8.9 (38.10) | 2.1 (31.05) | 0.8 (36.66)

21. Secondary Outcome: Change From Baseline to Week 2 in the Median Value for Actigraphy Data of Average Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in average activity per epoch (counts/epoch) to Week 2.
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | -15.4 (27.93) | -7.9 (38.40) | -7.2 (30.97) | 13.1 (40.32)

22. Secondary Outcome: Change From Baseline to Week 3 in the Median Value for Actigraphy Data of Average Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in average activity per epoch (counts/epoch) to Week 3.
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 1.5 (38.40) | 7.2 (29.11) | 9.9 (35.90) | -1.6 (25.68)

23. Secondary Outcome: Change From Baseline to Week 4 in the Median Value for Actigraphy Data of Average Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in average activity per epoch (counts/epoch) to Week 4.
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | -15.4 (27.06) | 9.0 (34.81) | -0.4 (39.18) | -18.7 (39.70)

24. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Median Value for Actigraphy Data of Maximum Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline in maximum activity to Endpoint.
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had at least one assessment by actigraphy after baseline
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -124.3 (235.16) | -73.2 (284.32) | 70.4 (191.11) | -5.9 (267.21)

25. Secondary Outcome: Change From Baseline to Week 1 in the Median Value for Actigraphy Data of Maximum Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 1 in maximum activity.
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -85.7 (312.58) | 14.8 (365.46) | 20.5 (436.62) | 6.2 (309.81)

26. Secondary Outcome: Change From Baseline to Week 2 in the Median Value for Actigraphy Data of Maximum Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 2 in maximum activity.
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | -152.7 (244.27) | -146.3 (291.42) | 11.8 (282.99) | -28.4 (288.45)

27. Secondary Outcome: Change From Baseline to Week 3 in the Median Value for Actigraphy Data of Maximum Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 3 in maximum activity.
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 1420.4 (345.81) | 1522.5 (558.66) | 1469.2 (440.96) | 1505.1 (356.41)

28. Secondary Outcome: Change From Baseline to Week 4 in the Median Value for Actigraphy Data of Maximum Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to week 4 in maximum activity.
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | -173.5 (371.31) | -61.4 (335.30) | 57.5 (218.02) | -60.4 (286.13)

29. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Median Value for Actigraphy Data of Standard Deviation of Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to endpoint in standard deviation of activity (counts/epoch).
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had at least one assessment by actigraphy after baseline
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -5.1 (17.97) | -0.7 (25.68) | 6.0 (17.04) | -1.9 (20.07)

30. Secondary Outcome: Change From Baseline to Week 1 in the Median Value for Actigraphy Data of Standard Deviation of Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 1 in standard deviation of activity (counts/epoch).
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -4.3 (20.75) | 7.6 (27.14) | 4.2 (23.35) | 1.7 (32.05)

31. Secondary Outcome: Change From Baseline to Week 2 in the Median Value for Actigraphy Data of Standard Deviation of Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 2 in standard deviation of activity (counts/epoch).
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | -11.3 (23.14) | -6.6 (31.61) | -6.6 (21.20) | -0.3 (24.53)

32. Secondary Outcome: Change From Baseline to Week 3 in the Median Value for Actigraphy Data of Standard Deviation of Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 3 in standard deviation of activity (counts/epoch).
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 5.2 (32.29) | -6.6 (29.58) | 15.2 (26.98) | 1.1 (26.70)

33. Secondary Outcome: Change From Baseline to Week 4 in the Median Value for Actigraphy Data of Standard Deviation of Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to week 4 in standard deviation of activity (counts/epoch).
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | -7.9 (26.27) | 6.3 (30.62) | 7.4 (40.16) | -7.6 (23.50)

34. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Median Value for Actigraphy Data of Total Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Endpoint in total activity.
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had at least one assessment by actigraphy after baseline
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | 7037.0 (63882.86) | -9164.8 (75454.69) | 23631.1 (70519.50) | -24811.4 (95900.22)

35. Secondary Outcome: Change From Baseline to Week 1 in the Median Value for Actigraphy Data of Total Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to week 1 in total activity.
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | 5913.6 (63868.75) | -3818.5 (78107.11) | 23665.1 (83030.07) | -12675.4 (118072.5)

36. Secondary Outcome: Change From Baseline to Week 2 in the Median Value for Actigraphy Data of Total Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 2 in total activity.
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | 2346.8 (45862.44) | -32082.8 (91836.83) | 3103.1 (69263.03) | 30660.0 (111626.4)

37. Secondary Outcome: Change From Baseline to Week 3 in the Median Value for Actigraphy Data of Total Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 3 in total activity.
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 39831.8 (115073.2) | 16850.4 (55047.52) | 56889.1 (83338.41) | 29067.5 (178423.5)

38. Secondary Outcome: Change From Baseline to Week 4 in the Median Value for Actigraphy Data of Total Activity
Description: An actigraphy device was worn by each patient starting with the initial screening. The device continuously measured movement, allowing for an evaluation of spontaneous motor activity. Data from the actigraphy device were downloaded at each visit. The data presented here is the change from baseline to Week 4 in total activity.
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | 1341.8 (92122.95) | 12620.9 (88874.07) | 55151.0 (67614.02) | -24323.9 (104375.7)

39. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Minimum Value for Actigraphy Data of Total Activity
Description: as for outcome 34
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had at least one assessment by actigraphy after baseline
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | -41210.0 (97542.44) | -16150.5 (45645.34) | -5159.5 (25855.48) | -34443.8 (72427.27)

40. Secondary Outcome: Change From Baseline to Week 1 in the Minimum Value for Actigraphy Data of Total Activity
Description: as for outcome 35
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | 2419.5 (147029.2) | 37665.8 (124537.9) | 15892.7 (36649.79) | 1116.3 (100205.7)

41. Secondary Outcome: Change From Baseline to Week 2 in the Minimum Value for Actigraphy Data of Total Activity
Description: as for outcome 36
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | -3534.2 (45509.04) | 27543.3 (89272.51) | 7937.0 (19889.36) | 27759.5 (100774.8)

42. Secondary Outcome: Change From Baseline to Week 3 in the Minimum Value for Actigraphy Data of Total Activity
Description: as for outcome 37
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 89886.7 (58766.65) | 91057.2 (105129.3) | 126496.5 (71256.20) | 60259.0 (81898.19)

43. Secondary Outcome: Change From Baseline to Week 4 in the Minimum Value for Actigraphy Data of Total Activity
Description: as for outcome 38
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | -12493.6 (40759.54) | -6742.8 (45841.91) | 39458.0 (36820.07) | 1744.3 (92667.31)

44. Other Pre Specified Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Modified Simpson-Angus Scale Total Score
Description: The Modified Simpson Angus Scale is a clinician-rated scale to assess the presence and severity of extrapyramidal symptoms associated study drug treatment. This is a 10-item scale that focuses on rigidity. The items are rated using a 5-point (0 - 4) scale. The total score ranges between 0 and 40. The data presented here represents the change from Baseline to Week 4 or the last observation following baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: Safety Analysis Set defined as subjects who had at least one dose of study medication and an observation at baseline and at least one observation after baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 14
Units on a scale | 0.1 (0.46) | -0.1 (1.33) | -0.3 (0.83) | 0.3 (0.61)

45. Other Pre Specified Outcome: Change From Baseline to Week 1 in the Modified Simpson-Angus Scale Total Score
Description: The Modified Simpson Angus Scale is a clinician-rated scale to assess the presence and severity of extrapyramidal symptoms associated study drug treatment. This is a 10-item scale that focuses on rigidity. The items are rated using a 5-point (0 - 4) scale. The total score ranges between 0 and 40. The data presented here represents the change from Baseline to Week 1.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose clinician completed an efficacy assessment at week 1. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 13 | 12 | 14
Units on a scale | 0.0 (0.38) | -0.2 (0.38) | -0.1 (1.00) | -0.1 (0.47)

46. Other Pre Specified Outcome: Change From Baseline to Week 2 in the Modified Simpson-Angus Scale Total Score
Description: The Modified Simpson Angus Scale is a clinician-rated scale to assess the presence and severity of extrapyramidal symptoms associated study drug treatment. This is a 10-item scale that focuses on rigidity. The items are rated using a 5-point (0 - 4) scale. The total score ranges between 0 and 40. The data presented here represents the change from Baseline to Week 2.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale | 0.1 (0.28) | -0.4 (2.23) | -0.3 (1.14) | 0.0 (0.41)

47. Other Pre Specified Outcome: Change From Baseline to Week 4 in the Modified Simpson-Angus Scale Total Score
Description: The Modified Simpson Angus Scale is a clinician-rated scale to assess the presence and severity of extrapyramidal symptoms associated study drug treatment. This is a 10-item scale that focuses on rigidity. The items are rated using a 5-point (0 - 4) scale. The total score ranges between 0 and 40. The data presented here represents the change from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose clinician completed an efficacy assessment at week 4. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
Units on a scale | -0.1 (0.29) | -0.1 (1.44) | -0.2 (0.72) | 0.2 (0.60)

48. Other Pre Specified Outcome: Change From Baseline to Week 4 or Last Observation Following Baseline in the Barnes Akathisia Scale (BARS) Total Score
Description: The BARS is a 4-item clinician-rated scale to measure the presence and severity of drug-induced akathisia. Items related to the assessment of objective akathisia, subjective awareness of restlessness, and distress related to restlessness are rated using various 4-point (0 - 3) scales. A global assessment of akathisia is rated using a 6-point (0=Absent, 1=Questionable akathisia, 2=Mild akathisia, 3=Moderate akathisia, 4=Marked akathisia, 5=Severe akathisia) scale. The total score range is from 0 to 14 with a higher score indicating more severe akathisia.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 14 | 14 | 14
Units on a scale | -0.3 (1.05) | -0.1 (0.53) | -0.1 (0.53) | -0.1 (1.07)

49. Other Pre Specified Outcome: Change From Baseline to Week 1 in the Barnes Akathisia Scale (BARS) Total Score
Description: as for outcome 48
Time Frame: Baseline and 1 week following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 13 | 12 | 14
Units on a scale | -0.4 (1.12) | -0.2 (0.55) | 0.0 (0.85) | 0.1 (0.66)

50. Other Pre Specified Outcome: Change From Baseline to Week 2 in the Barnes Akathisia Scale (BARS) Total Score
Description: as for outcome 48
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose clinician completed an efficacy assessment at week 2. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale | 0.2 (0.83) | 0.1 (1.08) | -0.3 (0.62) | 0.4 (1.71)

51. Other Pre Specified Outcome: Change From Baseline to Week 4 in the Barnes Akathisia Scale (BARS) Total Score
Description: as for outcome 48
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
Units on a scale | -0.1 (0.29) | -0.2 (0.58) | -0.2 (0.58) | -0.1 (1.12)

52. Other Pre Specified Outcome: Change From Baseline to Week 4 or Last Observation After Baseline on the Calgary Depression Scale for Schizophrenia (CDSS) Total Score
Description: The CDSS is a clinician-rated scale that assesses the level of depression in patients with schizophrenia. Each of the 9 items is scored on a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe). The total score range is 0 - 27. The data presented here represents the change from Baseline to Week 4 or the last observation following baseline in the total score.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 14 | 12 | 14
Units on a scale | 0.2 (2.14) | -0.4 (1.83) | 0.3 (2.19) | 0.1 (1.29)

53. Other Pre Specified Outcome: Change From Baseline to Week 2 on the Calgary Depression Scale for Schizophrenia (CDSS) Total Score
Description: The CDSS is a clinician-rated scale that assesses the level of depression in patients with schizophrenia. Each of the 9 items is scored on a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe). The total score range is 0 - 27. The data presented here represents the change from Baseline to Week 2 in the total score.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale | 0.7 (2.75) | -1.1 (1.93) | -0.8 (1.19) | 0.4 (1.26)

54. Other Pre Specified Outcome: Change From Baseline to Week 4 on the Calgary Depression Scale for Schizophrenia (CDSS) Total Score
Description: The CDSS is a clinician-rated scale that assesses the level of depression in patients with schizophrenia. Each of the 9 items is scored on a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe). The total score range is 0 - 27. The data presented here represents the change from Baseline to Week 4 in the total score.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
Units on a scale | 0.0 (2.26) | -0.6 (1.93) | 0.3 (2.19) | 0.2 (1.34)

55. Other Pre Specified Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Positive Scale score ranges from 7 to 49. The data here represents the change in Positive Rating Scale from Baseline to Endpoint.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 14 | 13 | 14
Units on a scale | -0.7 (2.05) | 0.1 (3.34) | -0.4 (2.69) | -0.9 (1.21)

56. Other Pre Specified Outcome: Change From Baseline to Week 1 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Positive Scale score ranges from 7 to 49. The data here represents the change in Positive Rating Scale from Baseline to Week 1.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 15 | 13 | 12 | 14
Units on a scale | 0.3 (1.71) | -0.1 (1.71) | 0.3 (2.50) | -0.6 (1.50)

57. Other Pre Specified Outcome: Change From Baseline to Week 2 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Positive Scale score ranges from 7 to 49. The data here represents the change in Positive Rating Scale from Baseline to Week 2.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale | -0.3 (1.65) | -1.1 (1.88) | 0.4 (2.19) | -0.9 (1.04)

58. Other Pre Specified Outcome: Change From Baseline to Week 4 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Positive Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Positive Scale score ranges from 7 to 49. The data here represents the change in Positive Rating Scale from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
Units on a scale | -0.7 (2.02) | -0.8 (2.41) | -0.6 (2.71) | -1.0 (1.22)

59. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Maximum Value for Actigraphy Data of Total Activity
Description: as for outcome 34
Time Frame: Baseline and Week 4 or last observation after baseline
Population: Full analysis set defined as subjects who had at least one assessment by actigraphy after baseline
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | 175906.8 (234098.9) | 45621.4 (112402.4) | 144855.3 (191836.4) | 38708.1 (132339.4)

60. Secondary Outcome: Change From Baseline to Week 1 in the Maximum Value for Actigraphy Data of Total Activity
Description: as for outcome 35
Time Frame: Baseline and Week 1
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 1
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 12
Counts | 92077.4 (260737.6) | -28961.9 (96313.45) | 18639.8 (95180.94) | -118038 (388177.5)

61. Secondary Outcome: Change From Baseline to Week 2 in the Maximum Value for Actigraphy Data of Total Activity
Description: as for outcome 36
Time Frame: Baseline and Week 2
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 2
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 12
Counts | -46326.7 (105330.1) | -44034.8 (120738.2) | -1954.7 (97046.14) | -78154.5 (367148.4)

62. Secondary Outcome: Change From Baseline to Week 3 in the Maximum Value for Actigraphy Data of Total Activity
Description: as for outcome 37
Time Frame: Baseline and Week 3
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 3
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
Counts | 40120.5 (151218.3) | 23748.0 (107713.9) | 61304.7 (158096.3) | -41751.7 (117072.2)

63. Secondary Outcome: Change From Baseline to Week 4 in the Maximum Value for Actigraphy Data of Total Activity
Description: as for outcome 38
Time Frame: Baseline and Week 4
Population: Full analysis set defined as subjects who had an assessment by actigraphy at baseline and at Week 4
Measure: Mean (Standard Deviation); unit: Counts
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 8 | 10 | 10 | 10
Counts | 7898.0 (71370.81) | -10300.1 (165816.5) | 123442.9 (168028.8) | -240840 (666800.6)

64. Secondary Outcome: Change From Baseline to Endpoint (Week 4 or Last Observation After Baseline) in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Scores
Description: The SCoRS is an 18-item interview based assessment covering all the cognitive domains in the MATRICS Consensus Cognitive Battery except social cognition. It is administered separately to the patient and an informant (family or friend) who are asked to rate the patient's level of difficulty in performing various cognitive functions on a 4-point scale (higher rating = greater impairment). They also complete a global assessment of cognitive function on a 1-10 scale. The interviewer factors in their own assessment on both the 18-items (Total Score) and the global assessment for the final score.
Time Frame: Baseline and Week 4 or last observation after baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 10 | 14 | 10 | 10
Units on a scale | -3.9 (7.87) | -0.7 (8.22) | -4.6 (6.19) | -3.1 (4.28)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil treatment in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the SCoRS Total score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.12, 95% CI 2-sided [-0.76 to 1.0]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 64, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.33, 95% CI 2-sided [-1.15 to 0.48]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 64, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.27, 95% CI 2-sided [-0.61 to 1.15]

65. Secondary Outcome: Change From Baseline to Week 2 in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Scores
Description: as for outcome 64
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had an efficacy assessment at week 2. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 10
Units on a scale | -5.0 (5.63) | -3.0 (6.88) | -1.6 (3.17) | -3.3 (4.16)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.33, 95% CI 2-sided [-0.58 to 1.24]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.05, 95% CI 2-sided [-0.91 to 0.81]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.44, 95% CI 2-sided [-1.33 to 0.45]

66. Secondary Outcome: Change From Baseline to Week 4 in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Scores
Description: as for outcome 64
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who had an efficacy assessment at week 4. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 9 | 11 | 10 | 9
Units on a scale | -3.8 (8.33) | -1.8 (8.90) | -4.6 (6.19) | -2.6 (4.16)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.18, 95% CI 2-sided [-0.75 to 1.10]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.10, 95% CI 2-sided [-0.98 to 0.78]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.37, 95% CI 2-sided [-0.54 to 1.27]

67. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Global Rating
Description: as for outcome 64
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose interviewers completed an efficacy assessment at least once after baseline. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | 0.3 (1.86) | -0.2 (1.37) | -0.3 (1.50) | -0.4 (1.73)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.38, 95% CI 2-sided [-1.14 to 0.38]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.13, 95% CI 2-sided [-0.89 to 0.63]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.05, 95% CI 2-sided [-0.84 to 0.73]

68. Secondary Outcome: Change From Baseline to Week 2 in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Global Rating
Description: n The SCoRS is an 18-item interview based assessment covering all the cognitive domains in the MATRICS Consensus Cognitive Battery except social cognition. It is administered separately to the patient and an informant (family or friend) who are asked to rate the patient's level of difficulty in performing various cognitive functions on a 4-point scale (higher rating = greater impairment). They also complete a global assessment of cognitive function on a 1-10 scale. The interviewer factors in their own assessment on both the 18-items (Total Score) and the global assessment for the final score.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose interviewers completed an efficacy assessment at week 2. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | 0.0 (1.86) | -0.3 (0.98) | 0.6 (2.02) | -0.8 (1.71)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.41, 95% CI 2-sided [-1.21 to 0.40]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.29, 95% CI 2-sided [-1.09 to 0.52]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.69, 95% CI 2-sided [-1.51 to 0.14]

69. Secondary Outcome: Change From Baseline to Week 4 in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Global Rating
Description: as for outcome 64
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and whose interviewers completed an efficacy assessment at week 4. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 11 | 12 | 12 | 12
Units on a scale | -0.1 (1.45) | -0.4 (1.38) | -0.3 (1.50) | -0.5 (1.78)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.24, 95% CI 2-sided [-1.06 to 0.58]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.05, 95% CI 2-sided [-0.85 to 0.75]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.10, 95% CI 2-sided [-0.90 to 0.70]

70. Secondary Outcome: Clinical Global Impression of Severity of Illness (CGI-S) Ratings at Week 4 or Last Observation Following Baseline
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The CGI-S was assessed at Baseline, Week 1, Week 2 and Week 4. Data is presented representing the number of subjects who rated each CGI-S score at Endpoint which is Week 4 or the last observation following Baseline.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: Full analysis set defined as the number of subjects who had at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Participants
  Normal | 0 | 0 | 0 | 0
  Borderline ill | 0 | 1 | 1 | 0
  Mildly ill | 11 | 8 | 10 | 11
  Moderately ill | 3 | 5 | 1 | 2
  Markedly ill | 0 | 0 | 0 | 0
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 0 | 0 | 0

71. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 4 or Last Observation Following Baseline
Description: The PGIC is a patient-rated scale of the change in disease severity. The PGIC uses the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. The number of subjects who rated each category at Week 4 or at the last observation following Baseline is presented.
Time Frame: Week 4 or last observation following Baseline
Population: Full analysis set defined as subjects who have at least one observation after Baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Participants
  Very much improved | 1 | 2 | 4 | 3
  Much improved | 3 | 2 | 1 | 2
  Minimally improved | 9 | 4 | 6 | 5
  No change | 0 | 5 | 0 | 2
  Minimally worse | 0 | 1 | 1 | 1
  Much worse | 1 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0

72. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in Scale for the Assessment of Negative Symptoms (SANS) Total Scores
Description: SANS is a clinician-rated instrument that rates the severity of negative symptoms of schizophrenia. It contains 25 items in 5 domains: affective flattening/blunting, alogia, avolition-apathy, anhedonia-asociality, attentional impairment. Items in a domain assess symptoms and a global item assesses the overall severity of the domain. Each item is scored on a 6-point severity scale(0=Not at all, 1=questionable decrease, 2=mild, 3=moderate, 4=marked, 5=severe). The total scale ranges from 0-125. Data presented here represents change in total score from Baseline to Endpoint.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: Full analysis set defined as the number of subjects who had at least one baseline observation and one observation after baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -5.6 (11.78) | -3.0 (9.77) | -7.4 (14.23) | -6.1 (9.78)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil treatment in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the SANS Total score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.05, 95% CI 2-sided [-0.80 to 0.71]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 72, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.31, 95% CI 2-sided [-1.06 to 0.45]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 72, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.11, 95% CI 2-sided [-0.68 to 0.89]

73. Secondary Outcome: Change From Baseline to Week 1 in Scale for the Assessment of Negative Symptoms (SANS) Total Scores
Description: SANS is a clinician-rated instrument that rates the severity of negative symptoms of schizophrenia. It contains 25 items in 5 domains: affective flattening/blunting, alogia, avolition-apathy, anhedonia-asociality, attentional impairment. Items in a domain assess symptoms and a global item assesses the overall severity of the domain. Each item is scored on a 6-point severity scale(0=Not at all, 1=questionable decrease, 2=mild, 3=moderate, 4=marked, 5=severe). The total scale ranges from 0-125. Data presented here represents change in total score from Baseline to Week 1.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Units on a scale | -1.4 (4.11) | -2.5 (7.62) | -2.2 (13.11) | -2.2 (6.73)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.13, 95% CI 2-sided [-0.88 to 0.63]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.05, 95% CI 2-sided [-0.72 to 0.82]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.00, 95% CI 2-sided [-0.80 to 0.81]

74. Secondary Outcome: Change From Baseline to Week 2 in Scale for the Assessment of Negative Symptoms (SANS) Total Scores
Description: SANS is a clinician-rated instrument that rates the severity of negative symptoms of schizophrenia. It contains 25 items in 5 domains: affective flattening/blunting, alogia, avolition-apathy, anhedonia-asociality, attentional impairment. Items in a domain assess symptoms and a global item assesses the overall severity of the domain. Each item is scored on a 6-point severity scale(0=Not at all, 1=questionable decrease, 2=mild, 3=moderate, 4=marked, 5=severe). The total scale ranges from 0-125. Data presented here represents change in total score from Baseline to Week 2.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | 0.4 (10.13) | -4.5 (12.08) | -4.4 (13.87) | -6.8 (12.11)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.62, 95% CI 2-sided [-1.44 to 0.20]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.18, 95% CI 2-sided [-0.98 to 0.62]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.17, 95% CI 2-sided [-0.97 to 0.63]

75. Secondary Outcome: Change From Baseline to Week 4 in Scale for the Assessment of Negative Symptoms (SANS) Total Scores
Description: SANS is a clinician-rated instrument that rates the severity of negative symptoms of schizophrenia. It contains 25 items in 5 domains: affective flattening/blunting, alogia, avolition-apathy, anhedonia-asociality, attentional impairment. Items in a domain assess symptoms and a global item assesses the overall severity of the domain. Each item is scored on a 6-point severity scale(0=Not at all, 1=questionable decrease, 2=mild, 3=moderate, 4=marked, 5=severe). The total scale ranges from 0-125. Data presented here represents change in total score from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -5.3 (12.73) | -5.6 (6.97) | -7.4 (14.23) | -6.3 (10.17)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.08, 95% CI 2-sided [-0.88 to 0.72]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.08, 95% CI 2-sided [-0.88 to 0.72]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.08, 95% CI 2-sided [-0.72 to 0.89]

76. Secondary Outcome: Change From Baseline to Week 4 or Last Observation After Baseline in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Negative Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Negative Scale score ranges from 7 to 49. The data here represents the change in Negative Rating Scale from Baseline to Endpoint.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -0.3 (4.03) | -0.3 (3.43) | -3.4 (2.07) | 0.1 (1.93)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the PANSS Negative Scale score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.11, 95% CI 2-sided [-0.65 to 0.87]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 76, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.13, 95% CI 2-sided [-0.63 to 0.88]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 76, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 1.69, 95% CI 2-sided [0.78 to 2.60]

77. Secondary Outcome: Change From Baseline to Week 1 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Negative Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Negative Scale score ranges from 7 to 49. The data here represents the change in Negative Rating Scale from Baseline to Week 1.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Units on a scale | 0.4 (2.71) | -0.1 (3.28) | -2.5 (1.97) | -0.4 (2.60)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.30, 95% CI 2-sided [-1.06 to 0.46]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.10, 95% CI 2-sided [-0.87 to 0.67]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.89, 95% CI 2-sided [0.05 to 1.74]

78. Secondary Outcome: Change From Baseline to Week 2 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Negative Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Negative Scale score ranges from 7 to 49. The data here represents the change in Negative Rating Scale from Baseline to Week 2.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -0.1 (3.18) | -1.4 (2.61) | -2.3 (2.05) | -0.8 (1.82)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.25, 95% CI 2-sided [-1.05 to 0.55]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.29, 95% CI 2-sided [-0.52 to 1.09]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.75, 95% CI 2-sided [-0.08 to 1.58]

79. Secondary Outcome: Change From Baseline to Week 4 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Negative Scale Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Negative Scale score ranges from 7 to 49. The data here represents the change in Negative Rating Scale from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -0.1 (4.29) | -1.3 (2.38) | -3.4 (2.07) | 0.0 (2.00)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.02, 95% CI 2-sided [-0.78 to 0.82]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.55, 95% CI 2-sided [-0.27 to 1.36]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 1.62, 95% CI 2-sided [0.70 to 2.55]

80. Secondary Outcome: Change From Baseline to Week 4 or Last Observation Following Baseline in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Total Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Total score ranges from 7 to 210. The data here represents the change in Total score from Baseline to Endpoint.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -2.5 (8.56) | -0.9 (7.77) | -6.3 (7.25) | -1.7 (4.89)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the PANSS Total score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.11, 95% CI 2-sided [-0.64 to 0.87]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 76, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.11, 95% CI 2-sided [-0.87 to 0.64]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 76, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.73, 95% CI 2-sided [-0.08 to 1.54]

81. Secondary Outcome: Change From Baseline to Week 1 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Total Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Total score ranges from 7 to 210. The data here represents the change in Total score from Baseline to Week 1.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Units on a scale | 0.5 (4.97) | -0.8 (4.82) | -4.0 (4.86) | -2.3 (5.92)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.50, 95% CI 2-sided [-1.27 to 0.27]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.28, 95% CI 2-sided [-1.05 to 0.50]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.30, 95% CI 2-sided [-0.51 to 1.11]

82. Secondary Outcome: Change From Baseline to Week 2 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Total Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Total score ranges from 7 to 210. The data here represents the change in Total score from Baseline to Week 2.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -2.1 (7.05) | -3.2 (5.15) | -3.0 (7.08) | -2.8 (4.32)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.12, 95% CI 2-sided [-0.92 to 0.68]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.07, 95% CI 2-sided [-0.73 to 0.87]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.03, 95% CI 2-sided [-0.77 to 0.83]

83. Secondary Outcome: Change From Baseline to Week 4 in the Positive and Negative Symptom Scale for Schizophrenia (PANSS) Total Score
Description: PANSS is a clinician-rated instrument that rates the severity of psychopathology in patients with schizophrenia. 7 items measure positive symptoms (eg. delusions, hallucinations), 7 items measure negative symptoms (eg. blunted affect, social withdrawal), 16 items form a General Psychopathology scale (eg. anxiety, motor retardation). Each item is scored on a 7-point severity scale: 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. The Total score ranges from 7 to 210. The data here represents the change in Total score from Baseline to Week 4.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -2.1 (7.39) | -3.1 (5.85) | -6.3 (7.25) | -2.1 (4.89)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.00, 95% CI 2-sided [-0.80 to 0.80]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.18, 95% CI 2-sided [-0.62 to 0.98]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.66, 95% CI 2-sided [-0.16 to 1.49]

84. Secondary Outcome: Change From Baseline to Week 4 or Last Observation Following Baseline in Epworth Sleepiness Scale (ESS) Total Scores
Description: ESS is a self-administered subjective measure of daytime sleepiness, based on responses to questions referring to 8 everyday situations (eg. sitting and reading, talking to someone) and reflects a patient's propensity to fall asleep in those situations. Score for the ESS range from 0 to 24 with higher scores indicating greater daytime sleepiness. Data here represents the change from Baseline to Endpoint (Week 4 or last observation following baseline) in the ESS total score.
Time Frame: Baseline and 4 weeks (or last observation after Baseline)
Population: as for outcome 72
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Units on a scale | -2.1 (4.87) | -0.6 (5.36) | 1.0 (4.43) | -0.5 (7.48)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; This study was not designed for hypothesis testing, but to gather information relative to the efficacy of armodafinil in improving cognitive impairments in patients with schizophrenia. Inferential statistics were not performed. Effect sizes and 95% confidence intervals of the effect sizes for the change from baseline in the ESS Total score are provided for each armodafinil treated group compared with placebo. Actual changes from baseline are summarized using descriptive statistics; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.25, 95% CI 2-sided [-0.51 to 1.01]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 84, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.03, 95% CI 2-sided [-0.73 to 0.78]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 84, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.23, 95% CI 2-sided [-1.01 to 0.56]

85. Secondary Outcome: Change From Baseline to Week 1 in Epworth Sleepiness Scale (ESS) Total Scores
Description: ESS is a self-administered subjective measure of daytime sleepiness, based on responses to questions referring to 8 everyday situations (eg. sitting and reading, talking to someone) and reflects a patient's propensity to fall asleep in those situations. Score for the ESS range from 0 to 24 with higher scores indicating greater daytime sleepiness. Data here represents the change from Baseline to Week 1 in the ESS total score.
Time Frame: Baseline and 1 week following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who completed an efficacy assessment at week 1. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Units on a scale | -2.2 (5.39) | -1.4 (6.05) | 0.0 (2.65) | -1.5 (6.16)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.11, 95% CI 2-sided [-0.64 to 0.87]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.02, 95% CI 2-sided [-0.79 to 0.74]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.30, 95% CI 2-sided [-1.11 to 0.50]

86. Secondary Outcome: Change From Baseline to Week 2 in Epworth Sleepiness Scale (ESS) Total Scores
Description: ESS is a self-administered subjective measure of daytime sleepiness, based on responses to questions referring to 8 everyday situations (eg. sitting and reading, talking to someone) and reflects a patient's propensity to fall asleep in those situations. Score for the ESS range from 0 to 24 with higher scores indicating greater daytime sleepiness. Data here represents the change from Baseline to Week 2 in the ESS total score.
Time Frame: Baseline and 2 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who completed an efficacy assessment at week 2. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -1.1 (6.27) | -1.6 (6.33) | 0.3 (3.14) | -2.1 (6.68)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.15, 95% CI 2-sided [-0.95 to 0.65]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.07, 95% CI 2-sided [-0.87 to 0.73]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.43, 95% CI 2-sided [-1.24 to 0.38]

87. Secondary Outcome: Change From Baseline to Week 4 in Epworth Sleepiness Scale (ESS) Total Scores
Description: ESS is a self-administered subjective measure of daytime sleepiness, based on responses to questions referring to 8 everyday situations (eg. sitting and reading, talking to someone) and reflects a patient's propensity to fall asleep in those situations. Score for the ESS range from 0 to 24 with higher scores indicating greater daytime sleepiness. Data here represents the change from Baseline to Week 4 in the ESS total score.
Time Frame: Baseline and 4 weeks following the start of study drug administration
Population: Full analysis set defined as subjects who received one or more doses of the study drug and who completed an efficacy assessment at week 4. Summary statistics are provided for the observed data only, missing data was not estimated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units on a scale | -2.0 (5.29) | -0.5 (5.78) | 1.0 (4.43) | -1.7 (6.36)
Statistical Analysis 1: Comparison: Armodafinil 50 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = 0.06, 95% CI 2-sided [-0.75 to 0.86]
Statistical Analysis 2: Comparison: Armodafinil 100 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.19, 95% CI 2-sided [-0.99 to 0.62]
Statistical Analysis 3: Comparison: Armodafinil 200 mg/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inferential statistics were not performed; Effect size = -0.47, 95% CI 2-sided [-1.28 to 0.34]

88. Secondary Outcome: Clinical Global Impression of Severity of Illness (CGI-S) Ratings at Week 1
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The CGI-S was assessed at Baseline, Week 1, Week 2 and Week 4. Data is presented representing the number of subjects who rated each CGI-S score at week 1.
Time Frame: Baseline and 1 week
Population: as for outcome 45
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Participants
  Normal | 0 | 0 | 0 | 0
  Borderline ill | 0 | 0 | 1 | 0
  Mildly ill | 10 | 11 | 8 | 11
  Moderately ill | 3 | 2 | 2 | 1
  Markedly ill | 1 | 0 | 0 | 1
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 0 | 0 | 0

89. Secondary Outcome: Clinical Global Impression of Severity of Illness (CGI-S) Ratings at Week 2
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The CGI-S was assessed at Baseline, Week 1, Week 2 and Week 4. Data is presented representing the number of subjects who rated each CGI-S score at week 2.
Time Frame: Baseline and 2 weeks
Population: as for outcome 50
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Normal | 0 | 0 | 0 | 0
  Borderline ill | 0 | 1 | 1 | 0
  Mildly ill | 9 | 8 | 10 | 11
  Moderately ill | 3 | 3 | 1 | 1
  Markedly ill | 0 | 0 | 0 | 0
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 0 | 0 | 0

90. Secondary Outcome: Clinical Global Impression of Severity of Illness (CGI-S) Ratings at Week 4
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The CGI-S was assessed at Baseline, Week 1, Week 2 and Week 4. Data is presented representing the number of subjects who rated each CGI-S score at week 4.
Time Frame: Baseline and 4 weeks
Population: as for outcome 47
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Normal | 0 | 0 | 0 | 0
  Borderline ill | 0 | 1 | 1 | 0
  Mildly ill | 10 | 8 | 10 | 11
  Moderately ill | 2 | 3 | 1 | 1
  Markedly ill | 0 | 0 | 0 | 0
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 0 | 0 | 0

91. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 1
Description: The PGIC is a patient-rated scale of the change in disease severity. The PGIC uses the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. The number of subjects who rated each category at Week 1 is presented here.
Time Frame: Week 1
Population: as for outcome 85
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 13 | 11 | 13
Participants
  Very much improved | 1 | 2 | 2 | 1
  Much improved | 1 | 1 | 1 | 3
  Minimally improved | 2 | 0 | 6 | 4
  No change | 9 | 10 | 2 | 4
  Minimally worse | 0 | 0 | 0 | 1
  Much worse | 1 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0

92. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 2
Description: The PGIC is a patient-rated scale of the change in disease severity. The PGIC uses the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. The number of subjects who rated each category at Week 2 is presented here.
Time Frame: Week 2
Population: as for outcome 86
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very much improved | 1 | 2 | 2 | 3
  Much improved | 3 | 1 | 3 | 4
  Minimally improved | 2 | 3 | 5 | 2
  No change | 5 | 6 | 2 | 3
  Minimally worse | 1 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0

93. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 4
Description: The PGIC is a patient-rated scale of the change in disease severity. The PGIC uses the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse. The number of subjects who rated each category at Week 4 is presented here.
Time Frame: Week 4
Population: as for outcome 87
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Very much improved | 1 | 2 | 4 | 3
  Much improved | 3 | 2 | 1 | 2
  Minimally improved | 7 | 4 | 6 | 5
  No change | 0 | 4 | 0 | 1
  Minimally worse | 0 | 0 | 1 | 1
  Much worse | 1 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0

94. Secondary Outcome: Clinical Global Impression of Severity of Illness (CGI-S) Ratings at Baseline
Description: The CGI-S is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The CGI-S was assessed at Baseline, Week 1, Week 2 and Week 4. Data is presented representing the number of subjects who rated each CGI-S score at Baseline.
Time Frame: Baseline
Population: Full analysis set defined as the number of subjects who had at least one observation after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Number analyzed (Participants) | 14 | 14 | 12 | 13
Participants
  Normal | 0 | 0 | 0 | 0
  Borderline ill | 0 | 0 | 1 | 0
  Mildly ill | 10 | 11 | 8 | 11
  Moderately ill | 4 | 3 | 3 | 2
  Markedly ill | 0 | 0 | 0 | 0
  Severely ill | 0 | 0 | 0 | 0
  Among the most extremely ill | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a six weeks beginning with the Screening period (1 week), 4 weeks double-blind treatment and 1 week follow up. For subjects who discontinued early the follow up period was defined as 7 days after the final study visit.
Arm/Group | Armodafinil 50 mg/Day | Armodafinil 100 mg/Day | Armodafinil 200 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 8/15 | 6/15 | 8/15 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 50 mg/Day (N=15) | Armodafinil 100 mg/Day (N=15) | Armodafinil 200 mg/Day (N=15) | Placebo (N=14)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 50 mg/Day (N=15) | Armodafinil 100 mg/Day (N=15) | Armodafinil 200 mg/Day (N=15) | Placebo (N=14)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine kinase increased (Investigations) | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1
Hostility (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Retrograde Ejaculation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days